CLINICAL TRIAL: NCT04770896
Title: A Phase III, Open-Label, Randomized Study of Atezolizumab With Lenvatinib or Sorafenib Versus Lenvatinib or Sorafenib Alone in Hepatocellular Carcinoma Previously Treated With Atezolizumab and Bevacizumab
Brief Title: A Study of Atezolizumab With Lenvatinib or Sorafenib Versus Lenvatinib or Sorafenib Alone in Hepatocellular Carcinoma Previously Treated With Atezolizumab and Bevacizumab
Acronym: IMbrave251
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO42541
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Unresectable Hepatocellular Carcinoma
MeSH Terms: interventions — atezolizumab; lenvatinib; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atezolizumab + Lenvatinib or Sorafenib (Experimental): Participants will receive atezolizumab plus lenvatinib or sorafenib. Treatment will continue until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab; Drug: Lenvatinib; Drug: Sorafenib
- Lenvatinib or Sorafenib (Active Comparator): Participants will receive lenvatinib or sorafenib. Treatment will continue until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: Lenvatinib; Drug: Sorafenib

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab will be administered by intravenous (IV) infusion at a fixed dose of 1200 mg on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Other Names: Tecentriq
  Arms: Atezolizumab + Lenvatinib or Sorafenib
Drug: Lenvatinib — Lenvatinib will be administered once daily by mouth each day of every 21-day study treatment cycle. Participants with a baseline body weight of < 60 kg will receive a daily dose of 8 mg. Participants with a baseline body weight of ≥ 60 kg will receive a daily dose of 12 mg.
Drug: Sorafenib — Sorafenib will be administered at a dose of 800 mg per day, i.e. two tablets of 200 mg swallowed by mouth twice daily (equivalent to a total daily dose of 800 mg) each day of every 21-day study treatment cycle.

SUMMARY:
This is a Phase III, open-label, multicenter, randomized, two-arm study designed to evaluate the efficacy and safety of atezolizumab plus either lenvatinib or sorafenib versus lenvatinib or sorafenib alone in participants with locally advanced or metastatic Hepatocellular Carcinoma (HCC) who have progressed on prior systemic treatment with atezolizumab plus bevacizumab combination.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic and/or unresectable HCC with diagnosis confirmed by histology/ cytology or clinically by American Association for the Study of Liver Diseases (AASLD) criteria in cirrhotic patients.
* Disease progression following prior atezolizumab plus bevacizumab combination treatment for HCC, for at least 4 consecutive treatment cycles, and 2 subsequent tumor assessments. It is required that at least 1 tumor assessment shows either stable disease (SD), partial response (PR), or complete response (CR).
* At least one measurable (per RECIST v1.1) target lesion that has not been previously treated with local therapy or, if the target lesion is within the field of previous local therapy, has subsequently progressed in accordance with RECIST v1.1.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1 within 7 days prior to randomization
* Child-Pugh class A within 7 days prior to randomization
* Adequate hematologic and end-organ function

Exclusion Criteria:

* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases.
* History of leptomeningeal disease
* History of hepatic encephalopathy, preceding 6 months, unresponsive to therapy within 3 days
* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
* History of malignancy other than HCC within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Randomization until death from any cause (approximately 42 months)
  Overall survival (OS) is defined as the time from randomization into the study to death from any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Randomization until the first occurrence of disease progression or death from any cause whichever occurs first (approximately 42 months)
  Progression free survival (PFS) is defined as the time from randomization into the study to the first occurrence of disease progression or death from any cause (whichever occurs first).
Confirmed Objective Response Rate (ORR) | Approximately 42 months
  Confirmed Objective Response Rate (ORR) is defined as the proportion of patients with a best response of either complete or partial response.
Time to Progression (TTP) | Randomization until the first occurrence of disease progression (approximately 42 months)
  Time to Progression (TTP) is defined as the time from randomization to the first occurrence of disease progression.
Duration of Response (DOR) | Time from the first occurrence of a confirmed documented objective response to disease progression or death from any cause whichever occurs first (approximately 42 months)
  Duration of Response (DOR) is defined as the time from the first occurrence of a documented confirmed objective response to disease progression or death from any cause (whichever occurs first).
Time to confirmed deterioration (TTCD) | Randomization to first deterioration maintained for two consecutive assessments, or one assessment followed by death from any cause wthin 3 weeks or 6 weeks (approximately 42 months)
  Time to confirmed deterioration (TTCD), of health-related quality of life (HRQoL), is defined as the time from randomization to first confirmed deterioration (decrease from baseline of ≥ 10 points) maintained for two consecutive assessments, or one assessment followed by death from any cause within 3 weeks (if Cycle 1-6) or 6 weeks (if after Cycle 6) in the following European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQC30) scales (separately): physical function, role function, and GHS/QoL.
Percentage of Participants With Adverse Events | Throughout study duration (approximately 42 months)
Percentage of Participants With Adverse Events for Combination Treatment, Adverse Events Related to Atezolizumab, and TKI-Related Adverse Events | Throughtout study (approximately 42 months)
Number of Participants With Anti-Drug Antibodies (ADAs) to Atezolizumab | Throughout study (approximately 42 months)
Serum Concentration of Atezolizumab | At pre-defined intervals from first administration of study drug to approximately 42 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (123):
- Austria (4):
  - Medizinische Universität Innsbruck, Innsbruck
  - Uniklinikum Salzburg, LKH, Salzburg
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Klinik Favoriten, Vienna
- Belgium (5):
  - AZ KLINA, Brasschaat
  - Hospital Erasme, Brussels
  - Cliniques Universitaires St-Luc, Brussels
  - UZ Leuven, Leuven
  - AZ Delta (Campus Rumbeke), Roeselare
- Brazil (6):
  - Hospital Felicio Rocho, Belo Horizonte, Minas Gerais
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina - CEPEN, Florianópolis, Santa Catarina
  - Clinicas Oncologicas Integradas - COI, Rio de Janeiro
  - Beneficencia Portuguesa de Sao Paulo, São Paulo
- Bulgaria (2):
  - Multiprofile Hospital for Active Treatment Uni Hospital, Panagyurishte
  - Complex Oncological Center - Plovdiv, EOOD, Plovdiv
- Canada (4):
  - Arthur J.E. Child Comprehensive Cancer Center-Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
- China (10):
  - Hunan Cancer Hospital, Changsha
  - Fujian Provincial Hospital, Fuzhou
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou
  - Nanfang Hospital, Southern Medical University, Guangzhou
  - Anhui Province Cancer Hospital, Hefei
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Nanjing
  - Zhongshan Hospital Fudan University, Shanghai
  - Renji Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Tianjin Cancer Hospital, Tianjin
- Costa Rica (2):
  - Clinica CIMCA, San José
  - ICIMED Instituto de Investigación en Ciencias Médicas, San José
- Clinical Hospital Centre Zagreb, Zagreb, Croatia
- AirForce Specialized Hospital, Cairo, Egypt
- Estonia (2):
  - North Estonia Medical Centre, Oncology and hematology Clinic, Tallinn
  - Tartu University Hospital, Tartu
- TAYS Radius rakennus, Tampere, Finland
- France (11):
  - CHU Grenoble Sud, Grenoble
  - CHRU de Lille - Hopital Claude Huriez, Lille
  - APHM, Marseille
  - CH Saint Eloi, Montpellier
  - CHU de Nantes - Hotel Dieu, Nantes
  - APHP - Hopital Saint Antoine, Paris
  - CHU Bordeaux, Pessac
  - Centre Eugene Marquis;Service d'oncologie, Rennes
  - CHU de Toulouse - Hôpital Rangueil, Toulouse
  - Hopitaux de Brabois - Gastro-Entereologie, Vandœuvre-lès-Nancy
  - Hopital Paul Brousse, Villejuif
- Germany (5):
  - Klinik Johann Wolfgang von Goethe Uni, Frankfurt
  - Med. Hochschule Hannover, Hanover
  - Uniklinik Mainz, Mainz
  - Universität Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
- Greece (2):
  - Laiko General Hospital Athen, Athens
  - Agioi Anargiroi Hospital of Kifissia, Nea Kifissia
- Israel (3):
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
- Italy (12):
  - Fondazione Pascale, Napoli, Campania
  - Azienda Osp Uni Seconda Università Degli Studi Di Napoli, Napoli, Campania
  - Ospedale del Mare, Napoli, Campania
  - A.O. S. Orsola Malpighi, Bologna, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Fondazione IRCCS Ospedale Maggiore Policlinico, Milan, Lombardy
  - Azienda Ospedaliera Ordine Mauriziano di Torino, Turin, Piedmont
  - A.O.U. Policlinico Paolo Giaccone, Palermo, Sicily
  - Azienda Ospedaliero-Universitaria Careggi, Florence, Tuscany
  - Azlenda Ospendaliero-Universitaria Pisana, Pisa, Tuscany
  - IRCCS Istituto Oncologico Veneto (IOV), Padua, Veneto
- Japan (10):
  - Fujita Health University Hospital, Aichi
  - National Cancer Center Hospital East, Chiba
  - Kurume University Hospital, Fukuoka
  - Hiroshima University Hospital, Hiroshima
  - Japanese Red Cross Society Himeji Hospital, Hyōgo
  - Yokohama City University Medical Center, Kanagawa
  - The University of Osaka Hospital, Osaka
  - Kindai University Hospital, Osaka
  - Jichi Medical University Hospital, Tochigi
  - Japanese Red Cross Musashino Hospital, Tokyo
- Malaysia (2):
  - Uni Malaya Medical Center, Kuala Lumpur, FED. Territory of Kuala Lumpur
  - Institute Kanser Negara (IKN), Putrajaya, FED. Territory of Kuala Lumpur
- Philippines (3):
  - Cebu Doctors' University Hospital, Cebu City
  - Makati Medical Center, Makati City
  - The Medical City, Pasig
- Russia (3):
  - FSBI "National Medical Research Center of Oncology N.N. Blokhin?, Moscow, Moscow Oblast
  - Moscow City Oncology Hospital #62, Moscow, Moscow Oblast
  - I.M.Sechenov First Moscow State Medical University (1st MSMU), Moskva, Moscow Oblast
- University Medical Center Ljubljana, Ljubljana, Slovenia
- South Korea (4):
  - National Cancer Center, Goyang-si
  - CHA Bundang Medical Center, Gyeonggi-do
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Spain (9):
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Complejo Hospitalario Universitario de Santiago (CHUS), Santiago de Compostela, LA Coruna
  - Clinica Universitaria de Navarra, Pamplona/iruña, Navarre
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Clinica Universidad de Navarra Madrid, Madrid
  - START Madrid. Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Universitario la Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (2):
  - Inselspital Bern Medizin Gastroenterologie, Bern
  - Universitätsspital Zürich Medizin Gastroenterologie, Zurich
- Taiwan (2):
  - Chi-Mei Medical Centre, Tainan
  - National Taiwan University Hospital, Zhongzheng Dist.
- Thailand (2):
  - Chulalongkorn Hospital, Bangkok
  - Faculty of Med. Siriraj Hosp., Bangkok
- Turkey (Türkiye) (7):
  - Memorial Ankara Hastanesi, Ankara
  - Medipol Mega Üniversite Hastanesi Göztepe, Ba?c?lar
  - Bakirkoy Dr. Sadi Konuk Egitim ve Arastirma Hastanesi, Tibbi Onkoloji, Bakirkoy / Istanbul
  - Uludag Uni Hospital, Bursa
  - Ac?badem Altunizade Hastanesi, Istanbul
  - Ege Uni Medical Faculty Hospital, Izmir
  - Hacettepe Uni Medical Faculty Hospital, Sihhiye/Ankara
- United Kingdom (7):
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Royal Free Hospital, London
  - King College Hospital NHS Foundation Trust, London
  - Hammersmith Hospital, London
  - Christie Hospital Nhs Trust, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing